CLINICAL TRIAL: NCT06315231
Title: Efficacy and Safety of Edaravone Dexborneol Sublingual Tablet for Post-stroke Cognitive Impairment in Patients With Acute Ischemic Stroke: a Multicenter, Randomized, Double-blind, Placebo-controlled, Exploratory Phase II Clinical Trial.
Brief Title: Edaravone Dexborneol Sublingual Tablet for the PSCI in Acute Ischemic Stroke Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0308-02-Y-2-201
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Post-stroke Cognitive Impairment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of edaravone dexborneol sublingual tablet (Experimental): Patients will receive edaravone dexborneol sublingual tablet twice daily of 24 weeks.
  Interventions: Drug: Edaravone dexborneol sublingual tablet
- Placebo (Placebo Comparator): Patients will receive placebo twice daily of 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone dexborneol sublingual tablet — Patients will receive one edaravone dexborneol sublingual tablet twice daily for 24 weeks
  Arms: Group of edaravone dexborneol sublingual tablet
Drug: Placebo — Patients will receive one placebo twice daily for 24 weeks
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, exploratory Phase II clinical trial.

The goal of this clinical trial is to assess the safety and efficacy of edaravone dexborneol sublingual tablets for post-stroke cognitive impairment in patients with acute ischemic stroke.

Participants will be required to receive 24 weeks treatment of edaravone dexborneol sublingual tablets or placebo during this study. The safety and efficacy endpoints will be compared in the patients with edaravone dexborneol sublingual tablets or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years and ≤ 80 years, male or female.
2. Diagnosed as ischemic stroke, no significant pre-stroke functional disability (mRS score ≤ 1prior to stroke onset).
3. The National Institutes of Stroke Scale score ≤ 20 points.
4. Time from onset to obtained informed consent form is within 7 days (including 7 days).
5. Presence of cognitive dysfunction at screening, i.e., MoCA scale score < 22.
6. Patients with good cognitive function prior to stroke, without significant cognitive dysfunction and dementia.
7. Education level: primary school or above, and can complete the cognitive function test required per investigator's judgement.
8. female subjects of childbearing potential and male subjects whose female partners are of childbearing potential must be willing to and use contraception during the study treatment and within 30 days after the last dose of study drug and have no plans to donate sperm or eggs; female subjects of childbearing potential will have a negative pregnancy test;
9. obtain voluntary signed informed consent from the patient or his/her legal representative approved by the Ethics Committee.

Exclusion Criteria:

1. Presence of intracranial hemorrhagic disease confirmed by brain imaging.
2. Severe disturbance of consciousness: NIHSS 1a level of consciousness item score > 1 point.
3. Transient ischemic attack (TIA).
4. Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 120 mmHg after blood pressure control.
5. Poorly controlled diabetes (fasting blood glucose >10mmol/L and/or HbA1c>8%).
6. Patients with contraindications to MRI imaging.
7. For subjects who are scheduled to undergo EEG examination, Patients with contraindications for EEG examination.
8. Presence of cognitive dysfunction prior to stroke assessed by informants, that is, the average score of Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE, 16-item version) during the screening period was ≥ 3.19 and the total score was ≥ 51.
9. Patients who have been diagnosed with severe mental disorders prior to stroke.
10. Severe limb hemiplegia and aphasia and significantly affect cognitive function assessment.
11. Patients have received the cognitive enhancers and other anti-dementia drugs within 1 month before the screening period, including but not limited to cholinesterase inhibitors (donepezil, rivastigmine, galantamine) and non-competitive N-methyl-D-aspartate (NMDA) receptor antagonists (memantine) and other drugs (such as mannitol sodium capsules, Ginkgo Biloba Extract Injection, Compound Ginkgo Biloba Tablets, oxiracetam, aniracetam, piracetam，nicergoline, Lecanemab, Donanemab, Aducanumab, etc. ).
12. Have been diagnosed with severe active liver disease, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc.; or ALT or AST > 2.0 × ULN.
13. Has been diagnosed with severe active kidney disease, renal insufficiency; or serum creatinine > 1.5 × ULN.
14. Thrombectomy or interventional therapy has been applied or planned after this episode.
15. History of malignancy; except for subjects with non-melanoma skin cancer (NMSC) that has been successfully treated and limited cervical cancer in situ. Subjects with a diagnosis of malignancy after enrollment may continue to participate in the study or not at the discretion of the investigator and at the discretion of the subject;
16. Suffering from a severe systemic disease with an expected survival period of <1 year;
17. hypersensitivity to dextran camphene, natural ice chips or edaravone or excipients (mannitol, copovidone, microcrystalline cellulose, cross-linked povidone, silicon dioxide, magnesium stearate);
18. pregnancy, lactation, and patients planning pregnancy;
19. history of major surgery within 4 weeks prior to enrollment;
20. participation in another clinical study within 30 days prior to randomization, or ongoing participation in another clinical study;
21. in the opinion of the investigator, not suitable for participation in this clinical study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Until follow up 26 weeks or early termination
  Adverse events (AE), treatment-related adverse events (TRAE), serious adverse events (SAE) in each group.
Number of discontinuation/withdrawal patients | Until follow up 26 weeks or early termination
  Discontinuation/withdrawal of patients in each group, including discontinuation due to adverse events.
The changes of the Vascular Dementia Assessment Scale-cognitive subscale (VaDAS-Cog) scores. | Until follow up 24 weeks
  The changes of the scores of the Vascular Dementia Assessment Scale-cognitive subscale (VaDAS-Cog) in each group after 24 weeks of treatment were compared with baseline. The minimum score is 0 and maximum score is 115 and the higher scores means the worse outcome.

SECONDARY OUTCOMES:
The incidence of Post Stroke Cognitive Impairment（PSCI ）in each group | Week 12 and Week 24
  The incidence of PSCI in each group at the 12th and 24th week of treatment, defined as Proportion of patients with MoCA score <22
The changes of Mini-Mental State Examination (MMSE) score | Week 12 and Week 24
  Mini-Mental State Examination (MMSE) at the 12th and 24th week of treatment (MMSE) score changes from baseline. The minimum score is 0 and maximum score is 30 and the higher scores means the better outcome.
The changes of Montreal Cognitive Assessment (MoCA) scale | Week 12 and Week 24
  Montreal Cognitive Assessment at the 12th and 24th week of treatment (MoCA) scale score changes from baseline. The minimum score is 0 and maximum score is 30 and the higher scores means the better outcome.
The changes of MoCA subscales | Week 12 and Week 24
  MoCA subscales (including visuospatial and execution) at the 12th and 24th week of treatment Function, naming, delayed recall, attention, language, abstraction, Orientation 7 subitems) from baseline. The minimum score is 0 and maximum score is 30 and the higher scores means the better outcome.
Modified Rankin Scale (mRS) scores | Week 12 and Week 24
  Modified Rankin Scale (mRS) scores at the 12th and 24th week of treatment. The minimum score is 0 and maximum score is 5 and the higher scores means the worse outcome.
The changes of National Institutes of Health Stroke Scale | Week 4 , Week 12 and Week 24
  National Institutes of Health Stroke Scale at the 4th,12th and 24th weeks of treatment (NIHSS) score changes from baseline. The minimum score is 0 and maximum score is 42 and the higher scores means the worse outcome.
The changes of the Vascular Dementia Assessment Scale-cognitive subscale (VaDAS-Cog) scores. | Week 12
  The changes of the scores of the Vascular Dementia Assessment Scale-cognitive subscale (VaDAS-Cog) in each group after 12 weeks of treatment were compared with baseline. The minimum score is 0 and maximum score is 115 and the higher scores means the worse outcome.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Taihe County People's Hospital, Fuyang, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Zhumadian Central Hospital, Zhumadian, Henan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Health Industry Group Bensteel General Hospital, Benxi, Liaoning
  - The First Hospital of Dalian Medical University, Dalian, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Tai'an Central Hospital, Taian, Shandong
  - Suining Central Hospital, Suining, Sichuan
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - The First People's Hospital of Huzhou, Huzhou, Zhejiang
  - Zhuji People's Hospital of Zhejiang Province, Zhuji, Zhejiang

IPD SHARING:
Plan to Share IPD: No